CLINICAL TRIAL: NCT06018818
Title: BIO|MASTER.Amvia: Post Market Clinical Follow-up Study for the Amvia/Solvia Pacemaker Family
Brief Title: Post Market Clinical Follow-up Study for the Amvia/Solvia Pacemaker Family
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biotronik SE & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BA114
Record Dates: First submitted 2023-07-17; First posted 2023-08-31 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-07

CONDITIONS: Bradycardia; Heart Failure
MeSH Terms: conditions — Bradycardia; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Amvia pacemaker or CRT-P implantation (Other)
  Interventions: Device: Amvia/Solvia pacemaker family

INTERVENTIONS:
Device: Amvia/Solvia pacemaker family — Implantation of a pacemaker or CRT-P devices

SUMMARY:
The study is designed as an open-label, prospective, international, multicenter, non-randomized study to determine safety and product performance of the CE-marked Amvia/Solvia pacemaker family, including the aATP, CRT AutoAdapt and Early Check features in the setting of a post-market clinical follow-up study.

ELIGIBILITY:
Inclusion Criteria:

* Standard indication for de novo, upgrade or replacement pacemaker or cardiac resynchronization therapy pacemaker (CRT-P) implantation
* Ability to understand the nature of the study
* Willingness to provide written informed consent
* Ability and willingness to perform all follow-up visits at the study site
* Ability and willingness to use the CardioMessenger and acceptance of the BIOTRONIK Home Monitoring® concept

Exclusion Criteria:

* Planned for conduction system pacing
* Planned cardiac surgical procedures or interventional measures other than the study procedure within the next 12 months
* Known pregnancy or breast feeding
* Age less than 18 years
* Participation in another interventional clinical investigation
* Life-expectancy less than 12 months

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2023-08-23 (Actual); Primary Completion 2025-07-21 (Actual); Study Completion 2025-07-21 (Actual)

PRIMARY OUTCOMES:
SADE-free rate at 6 months | 6 months
  Kaplan-Meier estimate of Amvia-related SADE-free rate at 6 months

SECONDARY OUTCOMES:
SADE-free rate at 12 months | 12 months
  Kaplan-Meier estimate of Amvia-related SADE-free rate at 12 months
CRT AutoAdapt performance | 12 months
  CRT AutoAdapt: different pacing percentages
CRT AutoAdapt AV delay | 12 months
  Mean adapted AV delay after pace/sense
Assessment of the CRT AutoAdapt feature (CRT-devices only) by the investigator | 12 months
  Investigator appraisal of the overall handling of the feature (score: very good/good/ adequate/poor/very poor)
Auto LV VectorOpt | 12 months
  Time needed for threshold measurement
Assessment of the Automatic LV VectorOpt test (CRT-devices only) by the investigator | 2 months
  Investigator appraisal of the overall handling of the feature (score: very good/good/ adequate/poor/very poor)
aATP-related ADEs and SADEs | 12 months
  aATP-related ADEs and SADEs
Sensing performance of device-based measurements | 12 months
  The appropriateness of sensing performance will be assessed by calculating the percentage of appropriate sensing for all leads.
Pacing performance of device-based measurements | 12 months
  The appropriateness of pacing performance will be assessed by calculating the percentage of appropriate pacing for all leads.

CONTACTS AND LOCATIONS:
Overall Officials: Istvan Szendey, Dr., Principal Investigator — Kliniken Maria Hilf GmbH
Locations (3):
- Kepler Universitätsklinikum, Linz, Austria
- Germany (2):
  - Elisabeth-Krankenhaus Essen, Essen
  - Kliniken Maria Hilf GmbH, Mönchengladbach

IPD SHARING:
Plan to Share IPD: No